CLINICAL TRIAL: NCT05382663
Title: Non-Invasive Monitoring of End-Stage Renal Disease Subjects Using Alio Medical Remote Monitoring System (RMS)
Brief Title: The Jordan Study for End-Stage Renal Disease Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AM14
Record Dates: First submitted 2022-04-02; First posted 2022-05-19 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ESKD Subjects (Experimental): Non-invasive device worn over vasculature.
  Interventions: Device: Alio Device

INTERVENTIONS:
Device: Alio Device — Non-invasive device worn over vasculature.

SUMMARY:
To compare the Alio device to blood draws.

DETAILED DESCRIPTION:
Eligible subjects who have signed a consent form will be asked to wear the Alio device at specified location(s) for up to four regularly scheduled dialysis sessions. The device will be placed and worn throughout the entire session.

Subjects will have blood draws that will be used to compare to device metrics. Additional vitals and monitoring may happen throughout this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* maintenance dialysis for ESRD via AVF/AVG in an arm location for at least 6 months
* written informed consent
* able to wear the SmartPatch as instructed and follow study protocols

Exclusion Criteria:

* Skin near the proximity of Patch placement is swollen, infected and/or inflamed
* pregnancy
* serious medical condition which in the opinion of the investigator may adversely affect the safety of the subject or the device being evaluated
* AVF/AVG in a non-arm location
* participants with novel indications for their AVG (ie. HeRO grafts)
* participation in any other clinical trials that could affect the quality of study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
1.Alio Device comparison to Hct via blood draw | through study completion, an average of 1 year
  Compare the Alio device to dialysis clinic blood lab values drawn before and after dialysis. The Hematrocrit (%) value collected will be compared to the Alio device.
1.Alio Device comparison to K+ via blood draw | through study completion, an average of 1 year
  Compare the Alio device to dialysis clinic blood lab values drawn before and after dialysis. The Potassium value collected will be compared to the Alio device.

CONTACTS AND LOCATIONS:
Overall Officials: Tawfiq Arafat, MD, Principal Investigator — Alkhansaa Hospital
Locations (1):
- Jordan Center for Pharmaceutical Research, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No